CLINICAL TRIAL: NCT00894270
Title: Comparison of Vehicle Delivery Depth Using the NovoFine® 5 mm Needle With or Without a Skin Fold and Inserted at Either 45 or 90 Degrees
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liggins Institute (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Paul Hofman/ Associate Professor, Liggins Institute, University of Auckland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Novofine002
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Injection; Needle
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sterile air injection — Injection of 20 microlitres using Novofine 5mm needle of sterile air into either abdomen or thigh using either a pinched or unpinched skin fold and either a vertical or angled approach.
Procedure: Placebo injection — Injection of either 20, 40 or 60 IU of placebo media into either abdomen or thigh using either a vertical or angled Novofine 5 mm needle. Leakage of fluid will be blotted and then weighed to establish fluid loss.
Device: Novofine needle — Novofine 5mm needle

SUMMARY:
Children and adolescents with type 1 diabetes mellitus are required to inject insulin daily. The injection technique should reliably deposit insulin into subcutaneous fat while minimizing inadvertent delivery into either the skin or the underlying muscle, both of which are associated with suboptimal outcomes. The use of shorter, thinner needles reduces the incidence of intramuscular delivery and is associated with reduced discomfort, but increases the risks of both shallow (intradermal) delivery and of loss of insulin through backflow to the skin surface.

In the current study, 240 subjects (children and adults) will receive multiple injections of small volumes of sterile air in the thigh and abdomen using 5 mm Novofine® needles, to simulate insulin injections performed at the two sites using various injection techniques (perpendicular or angled needle, with or without skin fold). Ultrasound visualisation of the injected air will allow determination of the incidence of intradermal or intramuscular delivery using the various delivery methods in the trial. In addition, adult subjects will receive injections of a liquid test medium in order to determine the incidence and extent of backflow. Qualitative data on perceived discomfort and information on body composition will also be collected. This investigation will form the basis for recommendations regarding preferred injection technique where 5 mm needles are used.

DETAILED DESCRIPTION:
Rationale:

The injection techniques used with children and adolescents with type 1 diabetes mellitus should reliably deposit insulin into subcutaneous fat while minimizing inadvertent intramuscular (IM) insulin injections. Surprisingly, injection technique varies among centres, tends to be protocol driven and is usually dependent on needle length. The recommended injection procedure for diabetic children in our centre include a lifted or pinched skin fold either on the abdomen, thigh or buttocks with perpendicular injection of 8 mm syringes and angled injection of 12.7 mm syringes. However both 8 and 12.7 mm needles, have been associated with frequent IM injections with rates of 38% and 86% respectively, reported using a perpendicular insertion (1, 2). IM injection of regular, NPH and glargine insulin has been associated with more rapid insulin release, variability in glycaemic control and an increased risk of hypoglycaemia (3-5).

The risk of IM insulin deposition is known to be related to a number of variables including younger age, male sex, lower body mass index (BMI), injection technique (angle of insertion and a lifted or pinched skinfold), and needle length (1, 2, 6-8). Reducing the length of the insulin needle reduces the incidence of IM injections, however the use of 5 mm insulin needles may result in insulin being administered too superficially in the dermal layer (9, 10). The consequence of intradermal insulin deposition is largely unknown, but may lead to increased insulin leakage, increased injection pain, and an increased immune response (10). Little information is known about skin thickness, although it does vary with age, obesity and puberty (personal observations).

Smaller, thinner needles are also associated with reduced pain and discomfort. However they may cause greater insulin loss after the injection. This latter issue may also reflect the injection technique used with anecdotal evidence suggesting angled techniques may reduce insulin loss.

Objectives:

Primary Objective: To locate and compare simulated insulin injections in children, adolescents and adults with diabetes given with 5 mm needle using a 45 degree and 90 degree injection angle, with and without skin fold in order to provide injection guidelines.

Secondary Objectives:

1. To study the thickness of dermis in abdomen and thigh in children, adolescents and adults with normal weight and over weight/obese.
2. To evaluate the distance from skin surface to muscle fascia (abdomen/thigh) with and without compression of the skin in children, adolescents and adults with normal weight and over weight/obese.
3. To quantify the amount of backflow of the test medium to the skin surface in adults and investigate whether there is a substantial clinically relevant difference among various techniques.
4. To assess comfort and ease of injection technique

This trial is a single-centre and open-label phase IV trial. The investigation will be performed in three visits. Patients screening will be done at the first visit, 2 ± 1 days prior to the second visit day. The second and the third visit will be performed with two weeks ± 3 days apart. At the second visit day all the subjects will receive (performed by study nurse) injected sterile air corresponding to 20 IU of insulin (200 µl) with Novofine 5 mm needles perpendicularly in abdomen and thigh with and without skin fold, giving in total four injections at this visit. Following the injection, sterile air deposition will be visualized by ultra sound (GELogic5 or a Phillips IU-22 machine). A 12.5 MHz linear array transducer will be used. This measures depth up to 3cm accurately. To assess dermis and air after injections a 1cm standoff will be employed. This is standard ultrasound technique to examine changes close to the transducer and we developed expertise using this technique during our previous study. Because of the better visualization using a standoff smaller, more physiological, volumes of air can be reliably injected. Thickness of (i) dermis and (ii) distance from skin surface to muscle fascia at the respective injection places will also be measured by ultrasound both with and without lifted skin fold prior to injection. The adults will be then injected with 200 µl of test medium with a 5 mm needle perpendicularly in abdomen and thigh with a lifted skin fold, providing an additional four injections to the adults. Possible backflow to skin surface will be absorbed by filter paper and quantified by scale. Injection speed will be measured by time from start to end of injection. After each injection subjects will be asked to complete a visual analog pain scale and after the injections they will be asked their preference for needle technique and site of injection. On the third visit day all subjects will be injected 200µl sterile air (performed by study nurse) with 5 mm needles at 45degrees with and without pinch-up technique in the abdomen and thigh, providing a total of four injections to each subject. In addition, 200µl test medium with 5 mm needle at 45degrees in abdomen and thigh with and without lifted skin fold will be injected to adults. Possible backflow to skin surface will be absorbed by filter paper and quantified by scale. The weighing scale must be able to measure with three decimals in the metric system (microgram). A 10 cm visual analog pain scale will be used to assess the discomfort of the injections in comparison to standard injections.

ELIGIBILITY:
Inclusion Criteria:

1. The subject/parent will give signed Informed Consent before any trial related activities. If the parents sign, it will be secured verbally or in older children in writing that they fully agree to participate.
2. Type 1 children aged ≥ 6 and < 19 years. Puberty will be determined by a trained paediatric endocrinologist using standard Tanner Staging.
3. Type 1 and 2 diabetic adults aged > 19 years and ≤ 85 years.

Exclusion Criteria:

1. Skin disease at abdomen and/or thigh.
2. Lipohypertrophy at the site of injection.
3. Any musculoskeletal abnormalities.
4. Psychiatric disorders.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Assess the safety and effectiveness of 5 mm needles using either thigh or abdomen and either a pinched or unpinched skin fold. | Assessed at the time of the injection

SECONDARY OUTCOMES:
Examine leakage of placebo medium from thigh or abdomen. | Immediately following the injection
Examine pain/discomfort of injections using the different techniques and the different injection sites. | Immediately following the injection

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Hofman, MD, Principal Investigator — Liggins Institute, University of Auckland
Locations (1):
- Liggins Institute, Auckland, Auckland, New Zealand

REFERENCES:
- [Background] Hofman PL, Lawton SA, Peart JM, Holt JA, Jefferies CA, Robinson E, Cutfield WS. An angled insertion technique using 6-mm needles markedly reduces the risk of intramuscular injections in children and adolescents. Diabet Med. 2007 Dec;24(12):1400-5. doi: 10.1111/j.1464-5491.2007.02272.x. PMID 18042081